CLINICAL TRIAL: NCT01044329
Title: Three Injections of Intravitreal Bevasizumab Versus Two Injections of Intravitreal Triamcinolone in the Management of Branch Retinal Vein Occlusion
Brief Title: Intravitreal Bevasizumab Versus Intravitreal Triamcinolone in Branch Retinal Vein Occlusion
Acronym: BRVO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Collaborators: Labbafinejad Medical Center (Other)
Responsible Party: Alireza ramezani, Ophthamic research center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8900
Record Dates: First submitted 2010-01-06; First posted 2010-01-07 (Estimated); Last update posted 2010-01-07 (Estimated); Status verified 2010-01

CONDITIONS: Branch Retinal Vein Occlusion
MeSH Terms: conditions — Retinal Vein Occlusion | interventions — Bevacizumab; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intravitreal bevacizumab (Active Comparator)
  Interventions: Drug: Bevacizumab
- Intravitreal triamcinolone (Active Comparator)
  Interventions: Drug: Triamcinolone Acetonide

INTERVENTIONS:
Drug: Bevacizumab — Intravitreal, 1.25 mg, 3 times, one month apart.
  Arms: Intravitreal bevacizumab
Drug: Triamcinolone Acetonide — Intravitreal, 2 mg, 2 times, two months apart.
  Arms: Intravitreal triamcinolone

SUMMARY:
This randomized clinical trial is conducted to evaluate the effect of three intravitreal injections of bevasizumab versus two intravitreal injections of triamcinolone in acute retinal vein occlusion. The outcomes are visual acuity and central macular thickness. The follow-up time is 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Recent onset (less than 3 months) BRVO

Exclusion Criteria:

* Any previous intervention

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-08 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Visual acuity | 6 months

SECONDARY OUTCOMES:
central macular thickness | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Imam Hossein medical center, Tehran, Iran